CLINICAL TRIAL: NCT05299333
Title: Comparison of the Effectiveness of Pulmonary Telerehabilitation and Physical Activity Recommendations in Patients With Pulmonary Fibrosis Due to COVID-19
Brief Title: Comparison of Pulmonary Telerehabilitation and Physical Activity Recommendations in Patients With Post Covid Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Ozge Ertan, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/25
Record Dates: First submitted 2022-03-25; First posted 2022-03-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Pulmonary Fibrosis
Keywords: Post covid fibrosis; Pulmonary Rehabilitation; Physical Activity
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): A total of 24 sessions of breathing exercises and high-repetitive muscle endurance and strengthening exercises will be applied to the pulmonary telerehabilitation group for 8 weeks, two days a week and one day a week unsupervised, via online systems. High-repetition muscle endurance and strengthening exercises will be applied to large muscle groups of the lower and upper extremities by creating resistance with body weight and theraband.
  Interventions: Other: Exercise
- Physical Activity Group (Active Comparator): Respiratory exercises and physical activity recommendations will be given to the physical activity group. Physical activity recommendations are; It will include information about the importance of physical activity and walking 3-5 days a week for at least 30 minutes of moderate intensity (4-6 on the Modified Borg scale of perceived exertion level).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — High repetition muscle endurance and strengthening exercises Walking

SUMMARY:
Rehabilitation plays a very important role in the management of patients with COVID-19, focusing on respiratory and motor functions, and therefore the importance of establishing treatment strategies to ensure optimal recovery of these patients has been emphasized. It has been stated that physical activity recommendations should be clarified for the management of symptoms associated with prolonged COVID-19 Syndrome and for the continuation of activities of daily living. It has been stated that after COVID-19 pneumonia, it is necessary to evaluate the physical functions of patients with long-term follow-up and to establish rehabilitation programs. The importance of being included in the rehabilitation program was emphasized, especially for patients with lung fibrosis.

The primary aim of this study was to compare the effects of pulmonary telerehabilitation and physical activity recommendations on exercise capacity and peripheral muscle strength in patients with pulmonary fibrosis due to COVID-19.

The secondary aim of this study is to compare the effects of pulmonary telerehabilitation and physical activity recommendations on symptoms, activity and participation in patients with pulmonary fibrosis due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients who have been infected with the COVID-19 virus at least three months ago and have been diagnosed with a positive PCR
* Patients with post-COVID-19 pulmonary fibrosis followed by a pulmonologist
* Patients who have sufficient technological infrastructure to participate in the telerehabilitation program and can adapt to online systems
* Patients who are clinically stable

Exclusion Criteria:

* Patients with orthopedic/neurological problems that prevent walking and exercise
* Patients with uncontrolled cardiovascular disease
* Patients with uncontrolled medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-04 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Submaximal exercise capacity | 1 week-8 week
  Six minute walk test and
maximal exercise capacity | 1 week-8 week
  Incremental shuttle walk test
endurance exercise capacity | 1 week-8 week
  endurance shuttle walk test
Peripheral muscle strength | 1 week-8 week
  Hand-held dynamometer

SECONDARY OUTCOMES:
Physical activity | 1 week-8 week
  Pedometer and activity monitor
Dyspnea | 1 week-8 week
  Modified Medical Research Council Dyspnea Scale stratifies severity of dyspnea in respiratory diseases. The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing
Fatigue | 1 week-8 week
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on patients. The FSS is a short questionnaire that requires to rate your level of fatigue. The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms. Patients read each statement and circle a number from 1 to 7, based on how accurately it reflects their condition during the past week and how much they agree or disagree that the statement applies to patients. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. Total score between 9-63. A total score of less than 36 suggests that you may not be suffering from fatigue.
Physical fitness | 1 week-8 week
  1 min sit to stand test
Functionality | 1 week-8 week
  Post covid-19 functionality scale (PCFS): The PCFS scale stratifies functional status limitation as follows: grade 0 (No functional limitations), grade 1 (Negligible functional limitations), grade 2 (Slight functional limitations), grade 3 (Moderate functional limitations), grade 4 (Severe functional limitations), and grade 5 (death)
System usability | 8 week
  System usability scale is a Likert Scale which includes 10 questions. Participants will rank each question from 1 to 5 based on how much they agree with the statement they are reading. 5 means they agree completely, 1 means they disagree vehemently.
Emotional status | 1 week-8 week
  Hospital anxiety and depression scale is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).
Body composition | 1 week-8 week
  Bioelectrical impedence analysis
Activities of daily living | 1 week-8 week
  London chest activity of daily living scale: Perceived dyspnea while performing daily living activities is scored between 0-5. A high score indicates greater disability in performing ADLs. The minimum score 0 and maximum total score is 75.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)